CLINICAL TRIAL: NCT05234112
Title: Prevention and Screening Intervention Project - Towards Elimination of Cervical Cancer
Brief Title: Prevention and Screening Towards Elimination of Cervical Cancer
Acronym: PRESCRIP-TEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Trnavska Universita v Trnavě (Unknown); Uganda Cancer Institute (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Manipal Academy for Higher Education (Unknown); Female Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202100943
Record Dates: First submitted 2022-01-03; First posted 2022-02-10 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: HPV Infection; Cervix Cancer; Cervical Dysplasia
Keywords: hrHPV test; screening cervical cancer; visual inspection cervix acetic acid; thermo-ablation; cryotherapy
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: In Uganda, India and Bangladesh eligible women in geographic areas are invited to perform self-test for hrHPV. hrHPV-positive women are invited for further examination of the cervix using VIA. In case of cervical dysplasia local treatment is performed.
  Women in vulnerable populations in Slovakia are invited to self-test for hrHPV. hrHPV positive women are seen by gynaecologist for Pap-smear cytology. Based on classification further therapy is offered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uganda, India, Bangladesh (Experimental): hrHPV self-test, followed by VIA inspection for hrHPV-positive women.
  Interventions: Behavioral: Community mobilisation for hrHPV self-testing; Diagnostic Test: hrHPV self-testing; Behavioral: Follow-up after testing; Diagnostic Test: VIA; Procedure: Thermo-ablation or cryotherapy for dysplasia
- Slovakia (Experimental): hrHPV self-test, followed by Pap-smear for cytology
  Interventions: Behavioral: Community mobilisation for hrHPV self-testing; Diagnostic Test: hrHPV self-testing; Behavioral: Follow-up after testing; Procedure: Thermo-ablation or cryotherapy for dysplasia; Diagnostic Test: Pap smear cytology

INTERVENTIONS:
Behavioral: Community mobilisation for hrHPV self-testing — use of social media, written media, theatre and other sources of communication to reach women, and relatives, to convince them of importance of screening.
Diagnostic Test: hrHPV self-testing — use of swabs that women insert in the vagina for taking sufficient material for testing for hrHPV. For women who are not confident to perform this this nurses provide assistance.
Behavioral: Follow-up after testing — based on the results of the test, follow-up is offered. In case of hrHPV negative test, retesting after five years. In case of hrHPV positive test, VIA in a nearby clinic. Women have to be motivated to adhere to follow-up
Diagnostic Test: VIA — Test offers insight into existence of dysplasia of the cervix by colouring the transition area
  Other Names: Visual Inspection of Cervix with Acetic Acid
  Arms: Uganda, India, Bangladesh
Procedure: Thermo-ablation or cryotherapy for dysplasia — Women with identified dysplasia lesions are offered immediate therapy to remove the infected superficial surface of the cervix
Diagnostic Test: Pap smear cytology — Cytology for identification of abnormal cells in the cervix, and classification of stages of dysplasia or pre-cancerous lesions
  Arms: Slovakia

SUMMARY:
The research project applies the protocol of the World Health Organisation for screening of cervical cancer, with testing of hrHPV as first screening, followed by Visual Inspection of the cervix with Acetic Acid for hrHPV-positive women and for women with minor lesions thermo-ablation of affected areas. This procedure is applied in Uganda, India and Bangladesh. In Slovakia hrHPV-positive women are offered Pap-smear and for women with Pap IV lis excision.

DETAILED DESCRIPTION:
The project performs community sensitisation and mobilisation in dedicated geographical areas and populations, to inform women and relatives about the importance of screening for cervical cancer.

To eligible women self-tests for hrHPV are offered, which can be applied at home and investigated in dedicated field-laboratories. Women who are hrHPV positive are invited for further diagnosis. In Uganda, India and Bangladesh Visual Inspection of the cervix with Acetic Acid is performed. In Slovakia Pap-smear. In case dysplasia is found, further treatment is performed with cryotherapy or thermo-ablation. Cases of suspect invasive cervical cancer are referred to hospitals for diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female in eligible age group
* Ability to give informed consent and participate in study

Exclusion Criteria:

* Clinical signs of cervical carcinoma
* Menstruation or other vaginal blood loss

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30000 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Uptake of hrHPV self-test in community | One week between approaching eligible women and collecting self-test
  Percentage of eligible women who take self-test out of women who have been offered self-test for hrHPV
Coverage of hrHPV self-test in community | 18 months between start approaching women in geographical area and closing screening operations in that area
  Percentage of women who take self-test out of women in geographical area eligible for self-test for hrHPV.
Uptake of VIA or Pap-smear of eligible women | One month between communicating hrHPV test result and measuring attendance in clinic for VIA or Pap-smear
  Percentage of women who are hrHPV-positive and are invited for VIA or Pap-smear who actually undergo the procedure

SECONDARY OUTCOMES:
Implementation fidelity of screening protocol | 24 months between start of preparations of health facilities for cervical cancer screening and measuring capabilities of health facility
  Percentage of health facilities involved in the research that is capable of performing the screening protocol fully (both human resources capacity as equipment and supplies
Sustainability of screening protocol | 24 months between start of preparations in geographical area and measuring cervical cancer screening policies and practices in organisation
  Percentage of local, district, regional health organisations involved in the study, that is able to maintain the screening protocol as Integrated part of service delivery

OTHER OUTCOMES:
Business case WHO screening protocol | 24 months between start data collection unit costs and production business case report
  Level of unit cost per screening following the new protocol and affordability in low and middle income countries

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Stekelenburg, PhD MD, Principal Investigator — University Medical Center Groningen; Janine de Zeeuw, PhD, Principal Investigator — University Medical Center Groningen; Martin Rusnak, PhD, Principal Investigator — Trnava University; Aminur Rahman Shaheen, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Carolyn Nakisige, MD, Principal Investigator — Uganda Cancer Institute; Shyamala Guruvare, PhD, Principal Investigator — Manipal Academy for Higher Education
Locations (1):
- Mpasana, Kakumiro, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Sharing according to the European Union Open Research guidelines
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 1 January 2024
Access Criteria: As per Open Research Protocol, on request to Principal Investigator UMCG
URL: http://www.prescriptec.org

REFERENCES:
- [Derived] Nazrul N, Rahman A, de Fouw M, Campbell C, Koot J, Kulsum MU, Ahmed MS, Haider SS, Hossain MA, Islam KM, Nessa A, Amrin M, Stekelenburg J, Beltman JJ. Cervical high-risk human papillomavirus infection and its associated risk factors: a community-based cross-sectional study in hard-to-reach areas in Bangladesh. BMJ Open. 2025 Dec 18;15(12):e103915. doi: 10.1136/bmjopen-2025-103915. PMID 41412622
- [Derived] Sultanov M, Zeeuw J, Koot J, der Schans JV, Beltman JJ, Fouw M, Majdan M, Rusnak M, Nazrul N, Rahman A, Nakisige C, Rao AP, Prasad K, Guruvare S, Biesma R, Versluis M, de Bock GH, Stekelenburg J. Investigating feasibility of 2021 WHO protocol for cervical cancer screening in underscreened populations: PREvention and SCReening Innovation Project Toward Elimination of Cervical Cancer (PRESCRIP-TEC). BMC Public Health. 2022 Jul 15;22(1):1356. doi: 10.1186/s12889-022-13488-z. PMID 35840949